CLINICAL TRIAL: NCT06813300
Title: Determination of Biomarkers of the Effectiveness of Deep Brain Stimulation by Direct Electrophysiological Recordings of Brain Activity in a Cognitive Context - LFP-DBS 2024
Acronym: LFP-DBS 2024
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D24-P005
Record Dates: First submitted 2024-09-24; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Pathology Requiring Deep Brain Stimulation Therapy
Keywords: DBS; LFP; MUA; MEG; IRM; cognitive tasks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive tasks performed during electrophysiological recordings (Experimental): Cognitive tasks performed during neural recordings (MUA, LFP) during the phases of a DBS
  Interventions: Procedure: Electrophysiological recordings

INTERVENTIONS:
Procedure: Electrophysiological recordings — Addition of electrophysiological recordings performed during cognitive tasks passation in patients undergoing DBS: in pre-op, per-op, peri-op and post-op setting

SUMMARY:
Deep brain stimulation (DBS) is a therapeutic approach aimed at applying high-frequency, low-intensity electrical stimulation using electrodes implanted in subcortical structures and connected subcutaneously to a stimulator implanted in the abdomen. In recent years, new indications have been studied for severe and drug-resistant forms of several neurological and neuropsychiatric pathologies. Its non-lesional, reversible and customizable nature make it a therapy of choice.

However, several factors are currently slowing down the evolution and optimization of SCP.

The identification of objective, quantifiable and predictive criteria for the therapeutic effects of stimulation would allow an acceleration of the individualized identification of the therapeutic parameters of SCP. The surgical procedure for implanting the stimulation equipment is carried out in several stages, which offer unique opportunities to acquire individual imaging or electrophysiology data that are potentially predictive of the therapeutic effect of DBS. In order to continue the optimization of DBS procedures, and therefore to maximize its therapeutic effects, it seems crucial to us to take advantage of all the neurophysiological data likely to be collected during this procedure. Furthermore, given the multiplication of indications for SCP, it seems necessary to highlight specific markers. Thus, the use of neurocognitive and/or motor tests specific to each pathology and coupled with electrophysiological recordings and anatomical and functional examinations would make it possible to highlight specific functional biomarkers predictive of therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient suffering from a pathology requiring treatment with deep brain stimulation: neurological disease (e.g.: Parkinson Disease, Essential Tremors, dystonia, epilepsy, etc.) or psychiatric disease (e.g.: Obsessive Compulsive Disorder, depression, eating disorders, etc.).
* Patient capable of understanding the study procedures and completing the self-questionnaires in French
* Patient informed and having signed the informed consent form

Exclusion Criteria:

* Contraindications to DBS, neurosurgery or anesthesia
* Patients with significant hemorrhagic or infectious risks
* Patient unable to perform the neurocognitive or sensorimotor tests
* Patient who is not a beneficiary of a social security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2036-04-25 (Estimated); Study Completion 2036-04-25 (Estimated)

PRIMARY OUTCOMES:
Brain activity recorded by electrophysiological measurements | From enrollment through study completion, an average of 2 years
  Electrophysiological variables recorded during neurocognitive and/or sensorimotor tests before and after the DBS procedure (at least 2 months at effective parameters)
Therapeutic effectiveness of DBS | From enrollment through study completion, , an average of 2 years
  The effectiveness of DBS is calculated as the differential (in %) of the symptom severity score(s) before and after the DBS procedure, measured using scales specific to each pathology (e.g. MADRS for depression (min score: 0 - max score: 60), YBOCS for OCD (min score: 0- max score: 40). Higher score means worse outcome for both scales.

SECONDARY OUTCOMES:
Number of patients with pre operative MRI by intensity | Day - 21
  Number of patients with 3 and 7 teslas MRI used before DBS surgery
Therapeutic effectiveness of DBS | From enrollment through study completion, an average of 2 years
  The effectiveness of DBS is calculated as the differential (in %) of the symptom severity score(s) before and after the DBS procedure, measured using scales specific to each pathology.
Number of participants with correct DBS electrodes implantation | Day 0
  The precision of the implantation of the DBS electrodes evaluated by the therapeutic effect obtained in the pathology treated.
Number of participants with inter-individual reproducibility of electrophysiological responses | From enrollment to the end of study at 18 months
  The inter-individual reproducibility of electrophysiological responses with a view to the generalization of this type of approach

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Grenoble-Alpes Hospital Center, Grenoble
  - Groupe Hospitalo-Universitaire Paris Psychiatrie et Neurosciences, Paris, Paris

IPD SHARING:
Plan to Share IPD: No